CLINICAL TRIAL: NCT02319928
Title: Randomized Controlled Trial of Comparison Between Surveillance Intervals After Excision of Colonic Adenomas
Brief Title: European Polyp Surveillance Trial
Acronym: EPoS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asociación Española de Gastroenterología (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AEG-EPOS-1
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short-term surveillance (Active Comparator): Short-term surveillance. Colonoscopy at 5+10 years in low-risk adenomas or 3+5 years in high-risk adenomas.
  Interventions: Procedure: Colonoscopy
- Long-term surveillance (Experimental): Long-term surveillance. Colonoscopy at 10 years in low-risk adenomas or 5 years in high-risk adenomas.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy

SUMMARY:
This protocol describes the epos (ancient greek (Επος) for "story") of a group of related clinical trials aiming at addressing one of the most important unsolved challenges in the prevention of colorectal cancer (one of our major cancer killers); the surveillance of patients with premalignant polyps in the large bowel.

This project is timely because large scale colorectal cancer screening programmes are currently rolled out in most Western countries. These programmes are diagnosing large numbers of individuals with premalignant polyps (adenomas and serrated polyps). This creates both a diagnostic and resource dilemma, because the optimal surveillance strategy for these individuals to reduce future cancer risk is currently unknown..

The EPoS trials will randomize or register more than 20,000 individuals in different European countries to different surveillance colonoscopy intervals to disentangle the most effective and cost-effective surveillance strategy for the population. Subjects will be randomized according to their presenting polyp chracteristics The EPoS I trial randomizes patients with low-risk adenomas into 5 or 10-year surveillance; ; EPoS II randomizes patients with high-risk adenomas into 3 or 5-yearly surveillance ; EPoS III will include patients with serrated polyps in a one-arm study with surveillance after 5 and 10 years. The primary endpoint for all three trials is incidence of colorectal cancer after 10 years of follow-up.

This EPoS trials are the largest in polyp surveillance ever conducted. They address a clinical problem affecting hundreds of thousand individuals in Europe and the US each year, it has a large size, and should thus provide definitive results.

ELIGIBILITY:
Inclusion Criteria:

* Cecal intubation (preferably documented by images/videoof the apendiceal orifice and the ileocecal valve; but not required).
* Adequate colonic cleansing, with Boston Bowel Cleansing Score equal or higher than 2 points in all colonic segments.
* Complete excision of all polyps at baseline colonoscopy findings (as judged by the trial endoscopists).

Exclusion Criteria:

* Lack of consent
* History of CRC or adenomas
* History of serrated polyps ≥ 10 mm in diameter at any colorectal location or ≥ 5 mm if located proximal to the splenic flexure
* Incomplete colonoscopy
* Incomplete endoscopic excision of polyps
* Genetic cancer syndrome (adenomatous or serrated polyposis syndrome; Lynch or Lynch-like syndrome)
* Inflammatory bowel disease
* History of surgical colon resection for any reason
* Severe co-morbidity with reduced life expectancy (NYHA 3-4)
* On-going cytotoxic treatment or radiotherapy for malignant disease
* Long-lasting attention and nursing services (somatic or psychosocial, mental retardation).

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2015-06; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer incidence | 10 years
  development of new colorectal cancer cases in the different arms of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Jover, MD, Principal Investigator — Hospital General Universitario de Alicante; Michael Bretthauer, MD, Principal Investigator — University of Oslo
Locations (1):
- Hospital General Universitario de Alicante, Alicante, Spain

REFERENCES:
- [Derived] Juul FE, Garborg K, Nesbakken E, Loberg M, Wieszczy P, Cubiella J, Kalager M, Kaminski MF, Erichsen R, Adami HO, Ferlitsch M, Furholm SKB, Zauber AG, Quintero E, Bugajski M, Holme O, Dekker E, Jover R, Bretthauer M. Rates of repeated colonoscopies to clean the colon from low-risk and high-risk adenomas: results from the EPoS trials. Gut. 2023 May;72(5):951-957. doi: 10.1136/gutjnl-2022-327696. Epub 2022 Oct 28. PMID 36307178
- [Derived] Jover R, Bretthauer M, Dekker E, Holme O, Kaminski MF, Loberg M, Zauber AG, Hernan MA, Lansdorp-Vogelaar I, Sunde A, McFadden E, Castells A, Regula J, Quintero E, Pellise M, Senore C, Kalager M, Dinis-Ribeiro M, Emilsson L, Ransohoff DF, Hoff G, Adami HO. Rationale and design of the European Polyp Surveillance (EPoS) trials. Endoscopy. 2016 Jun;48(6):571-8. doi: 10.1055/s-0042-104116. Epub 2016 Apr 4. PMID 27042931